CLINICAL TRIAL: NCT04714476
Title: Explorative, Monocentric, Feasibility Study Focusing on Fit of Innovative, Made-to-measure Compression Garments in Healthy Subjects II
Brief Title: Feasibility Study Focusing on Fit of Made-to-measure Compression Garments in Healthy Subjects II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BSN Medical GmbH (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BSN-C2673
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2021-01

CONDITIONS: Product Use Issue

STUDY DESIGN:
Intervention Model Description: Healthy subjects will test made-to-measure compression garments. No comparator group due to explorative design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fit test of made-to-measure garments (Experimental): Healthy subjects will test made-to-measure compression garments
  Interventions: Device: Made-to-measure compression garment

INTERVENTIONS:
Device: Made-to-measure compression garment — Subjects will wear one of two made-to-measure compression garments:
  (1) JOBST® Confidence leggins (BT) and (2) JOBST® Confidence Bermuda (ET)

SUMMARY:
Fit of made-to-measure compression garments in healthy subjects will be tested on one day, simulating daily activities.

DETAILED DESCRIPTION:
Lower extremities of 36 healthy subjects will be measured by trained experts to collect measures for made-to-measure compression garments.

Fit of made-to-measure compression garments, which are not on the market yet, among healthy subjects will be tested on one day, simulating daily activities. Fit will be assessed directly after donning and after a wearing period of maximum 7 hours at the study site by trained experts. Healthy subjects will give back study products at the end of the wearing period. AEs will be documented throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Men, women or diverse
* Full legal competence
* Age between 18 and 70 years
* Capability to understand the subject information and to provide conscious informed consent
* All female or diverse subjects of childbearing potential must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of a Pearl-Index less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices, sexual abstinence or vasectomized partner for at least 4 weeks
* Willingness to conduct a urine pregnancy test for all female or diverse subjects of childbearing potential
* Capability and willingness to follow protocol requirements
* Signed informed consent for study participation and data protection regulations
* BMI >23 kg/m² and ≤ 40 kg/m²

Exclusion Criteria:

* Circumference of the largest circumference of the upper leg >90 cm (measured in the upright position)
* Shape distortions between the waist and the feet
* Diagnosed lymphedema of the lower extremities
* Diagnosed lipedema of lower extremities
* Diagnosed indication for therapy with flat-knitted compression garments
* Alcohol abuse as reported by subject and/ or suspected by investigator
* Drug abuse as reported by subject and/ or suspected by investigator
* Allergy or sensitivity to one or more components of the investigational devices, as far as reported by the subject
* Pregnancy or breastfeeding
* Diagnosed peripheral arterial disease
* Presence of untreated phlebitis, or septic phlebitis
* Diagnosed progressed arterial insufficiency including ischemia
* Diagnosed congestive heart failure
* Diagnosed clinically relevant hypertension
* Diagnosed renal insufficiency or kidney failure
* Presence of Untreated or progressing skin infection
* Presence of large coagulum in the leg vein
* Presence of phlegmasia coerulea dolens
* Diagnosed Raynaud's disease
* Diagnosed gonarthrosis
* Diagnosed ankle arthrosis
* Diagnosed rheumatoid arthritis
* Presence of exuding dermatoses
* Presence of gangrene
* Diagnosed malign lymphedema
* Diagnosed psoriasis
* Diagnosed diabetes mellitus
* Diagnosed complex regional pain syndrome (CRPS; Sudeck atrophy)
* Diagnosed polyneuropathy
* Diagnosed severe impaired skin sensitivity und impaired sensitivity of the extremities, including all sensory malfunctions and diagnosed impaired pain sensitivity
* Objections of the investigator to the subject's participation in the trial due to medical reasons or any other reason for which the subject should not participate in the opinion of the investigator
* Participation in any clinical investigation with systemic and/or pharmaceutical substances within the last 4 weeks and/or in parallel
* Sponsors, manufacturers or CRO staff
* Surgery in the test area within the last 4 weeks
* Open wounds in the test area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the fit of the investigational device | One day
  Evaluation of the fit of the investigational medical device at the end of a wearing period of approximately 4 - 7 hours, to be worn by healthy subjects once.
  The fit will be evaluated visually as well as manually by predefined criteria, e.g. fit of the upper hem, fit of the investigational medical device at the body area, fit at the thighs, fit in the knee area, fit at the lower hem.
  The fit will be evaluated using a Visual Analog Scale VAS-10 (0=very good to 10= worse).

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, Dr., Principal Investigator — proDERM GmbH Institut für Angewandte Dermatologische Forschung
Locations (1):
- proDERM GmbH Institut für Angewandte Dermatologische Forschung, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. Data are needed for confidential medical device development.